CLINICAL TRIAL: NCT06012409
Title: Evaluation of the Occlusal Effects of the Hall Technique and Investigation of Children's Satisfaction
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Cardiff University (Other)
Responsible Party: Principal Investigator, Melis AKYILDIZ, Principle investigator, Aydin Adnan Menderes University
Other Study IDs: DHF-21008
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Dental Caries in Children
Keywords: Dental Caries; Children; Occlusion
MeSH Terms: conditions — Dental Caries; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hall Technique Prefabricated Metal Crown — The Hall Technique is a type of minimally invasive dental treatment. Hall Technique involves sealing the carious lesion under a Prefabricated Metal Crown to stop its progression preventing pain and/or infection.This makes the technique less invasive and it can be more acceptable to children than a traditional filling involving injections and drilling.

SUMMARY:
Background: The Hall Technique (HT) is a non-invasive, easily applicable minimally invasive dentistry approach for managing dental caries in children. It involves placing a preformed metal crown over a tooth with decay, to seal it in and stop the decay from progressing. However, it alters the occlusion as no tooth substance is removed to make space for the crown.

Objective: This study, aims to evaluate the effects of Hall Technique on occlusion in children, to assess whether there are any adverse effects on the temporomandibular joint and masseter muscles, related to changes on occlusion and to evaluate the children's perceptions of the crowns.

Materials and Methods: A total of 37 children aged 5-9 years, who have not been treated with the Hall Technique previously and who have dentinal caries that did not reach the pulp (affecting the occlusal or the occluso-proximal surfaces) in their primary molars, will be invited to participate in the study. At the first visit, clinical examination will be carried out and intraoral impressions will be taken for pre-treatment evaluation. The occlusal vertical dimension of the teeth will be measured clinically with callipers. Temporomandibular joint and masseter muscles will be examined clinically. Then, the Hall Technique crown will be placed to treat the carious tooth, the impressions taken again, and measurements repeated. At one and three months following treatment with the crown, the participant will have the measurements repeated. The child and parent will complete a questionnaire after 3 months on their perception of the crown.

In the data analysis, frequency, percentage, mean and standard deviation analyses will be used for demographic data and description of the clinical data. In numerical data analysis, t-test or Mann-Whitney U test will be used according to the data distribution. Geomagic software will be used to analyse sequential study models of the teeth to measure relative changes in the tooth positions over time.

DETAILED DESCRIPTION:
Dental caries is one of the most common chronic diseases during childhood. Due to the high incidence of dental caries in the primary dentition and inadequate treatments, early childhood caries is an important public health problem for children. The main challenge in paediatric dentistry, both for the clinician and the family, is to cooperate with the child to provide the necessary treatment successfully. Although many factors affect dental anxiety, research shows that the type of dental treatment can influence the child's behaviour. Minimally invasive dental approaches have been found to offer a more comfortable treatment process. The Hall Technique is a type of minimally invasive dental treatment. It has been used for more than 20 years to treat dental caries in children. In this technique, the carious lesion is sealed under a PMC to stop the progression of caries and prevent pain and/or infection. A crown is pressed over the tooth without local anaesthesia, tooth preparation/reduction, or carious tissue removal. This makes the technique less invasive and it can be more acceptable to children than a traditional filling involving injections and drilling.

One of the drawbacks of Hall Technique is that it increases the occlusal vertical dimension (OVD) because the PMC is placed on the tooth without any preparation. It is possible that an increase in the occlusal vertical dimension could cause hyperactivity of the masticatory muscles, an increase in occlusal forces, bruxism, and temporomandibular joint disorders. The Hall Technique has reportedly temporarily increased the vertical dimension. According to clinical research, it takes approximately a month for the vertical dimension to return its pre-treatment state.

To the best of our knowledge, none of the studies have accurately determined how the child's occlusion returns to its pre-treatment state after the placement of a Hall Technique preformed metal crown. The aim of this study is to evaluate the effects of Hall Technique on occlusion, temporomandibular joint, and masseter muscle in children and the child's perceptions of the crown.

ELIGIBILITY:
Children are eligible for inclusion if:

* they are 5 to 9 years old;
* they fit the clinical criteria to receive a HTPMC to manage primary molars carious lesions;
* they have antagonist primary molar
* they have not had a HTPMC fitted before;
* their parents can understand what is involved in the study and have signed and given assent to participate;
* they can cooperate with dental care including having a dental impression taken; and
* their parents are willing and able to bring them to the follow-up appointments 4, and 12 weeks after the treatment.

Children will be excluded from the study if:

* They do not have a parental agreement to participate; or
* They have self-reported occlusal parafunctional habits (e.g. bruxism, constantly open mouths).

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Potential participants will be selected and recruited from children attending for routine dental care at Aydin Adnan Menderes University Paediatric Dentistry Clinic.
  Children and their parents will be invited to participate and will be included in the study after they have the study discussed with them and they agree to participate, giving informed consent. Children should meet the inclusion criteria, and/or be none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Digital Occlusal Analysis | Baseline
  3D occlusal analysis will be performed on models taken from impressions of participants' teeth to evaluate the effects of the placement of a HTPMC on the occlusion (crowned teeth and the surrounding and opposing teeth).
Digital Occlusal Analysis | Immediately After Treatment
  3D occlusal analysis will be performed on models taken from impressions of participants' teeth to evaluate the effects of the placement of a HTPMC on the occlusion (crowned teeth and the surrounding and opposing teeth).
Digital Occlusal Analysis | 1 Month
  3D occlusal analysis will be performed on models taken from impressions of participants' teeth to evaluate the effects of the placement of a HTPMC on the occlusion (crowned teeth and the surrounding and opposing teeth).
Digital Occlusal Analysis | 3 Month
  3D occlusal analysis will be performed on models taken from impressions of participants' teeth to evaluate the effects of the placement of a HTPMC on the occlusion (crowned teeth and the surrounding and opposing teeth).

SECONDARY OUTCOMES:
Occlusal Vertical Dimension (OVD) Measurements | Baseline
  In order to determine whether OVD returns to pre-HTPMC placement levels, the occlusal vertical distance between the most prominent incisal points of the maxillary and mandibular cuspid/canine (on the same side of the jaw as that where the treatment takes place) will be scored. This will be measured in mm (from -10mm to 10mm) with a higher score indicating a worse outcome.
Occlusal Vertical Dimension (OVD) Measurements | Immediately After Treatment
  In order to determine whether OVD returns to pre-HTPMC placement levels, the occlusal vertical distance between the most prominent incisal points of the maxillary and mandibular cuspid/canine (on the same side of the jaw as that where the treatment takes place) will be scored.This will be measured in mm (from -10mm to 10mm) with a higher score indicating a worse outcome.This will be measured in mm (from -10mm to 10mm) with a higher score indicating a worse outcome.
Occlusal Vertical Dimension (OVD) Measurements | 1 month
  In order to determine whether OVD returns to pre-HTPMC placement levels, the occlusal vertical distance between the most prominent incisal points of the maxillary and mandibular cuspid/canine (on the same side of the jaw as that where the treatment takes place) will be scored. This will be measured in mm (from -10mm to 10mm) with a higher score indicating a worse outcome.
Occlusal Vertical Dimension (OVD) Measurements | 3 month
  In order to determine whether OVD returns to pre-HTPMC placement levels, the occlusal vertical distance between the most prominent incisal points of the maxillary and mandibular cuspid/canine (on the same side of the jaw as that where the treatment takes place) will be scored. This will be measured in mm (from -10mm to 10mm) with a higher score indicating a worse outcome.
Detect any negative effects on the TMJ | Baseline
  Clinical examination of the TMJ will be done according to AAPD Guidelines. The following questionnaire will be administered to children and parents to detect any negative effects. Does he/she have difficulty opening his/her mouth? a) Yes b) No Do you hear sounds inside your jaw joint? a) Yes b) No Is there pain in the ears or cheeks? a) Yes b) No Is there pain in the jaw when chewing, talking?
  a) Yes b) No Is there pain when chewing, talking?
  a) Yes b) No Is there pain when opening your mouth wide or yawning?
  a) Yes b) No Does biting feel uncomfortable or different from normal?
  a) Yes b) No Have you ever had locking or dislocation of the jaw?
  a) Yes b) No Is there a history of jaw, head or neck injury?
  a) Yes b) No If yes, when? How was it treated? Has he/she ever been treated for a jaw joint disorder?
  a) Yes b) No If so, when? How was it treated? Yes indicates a worse outcome
Detect any negative effects on the TMJ | Immediately after treatment
  Clinical examination of the TMJ will be done according to AAPD Guidelines.The following questionnaire will be administered to children and parents to detect any negative effects.Does he/she have difficulty opening his/her mouth? a) Yes b) No Do you hear sounds inside your jaw joint? a) Yes b) No Is there pain in the ears or cheeks? a) Yes b) No Is there pain in the jaw when chewing, talking?
  a) Yes b) No Is there pain when chewing, talking?
  a) Yes b) No Is there pain when opening your mouth wide or yawning?
  a) Yes b) No Does biting feel uncomfortable or different from normal?
  a) Yes b) No Have you ever had locking or dislocation of the jaw?
  a) Yes b) No Is there a history of jaw, head or neck injury?
  a) Yes b) No If yes, when? How was it treated? Has he/she ever been treated for a jaw joint disorder?
  a) Yes b) No If so, when? How was it treated? Yes indicates a worse outcome
Detect any negative effects on the TMJ | 1 month
  Clinical examination of the TMJ will be done according to AAPD Guidelines The following questionnaire will be administered to children and parents to detect any negative effects.Does he/she have difficulty opening his/her mouth? a) Yes b) No Do you hear sounds inside your jaw joint? a) Yes b) No Is there pain in the ears or cheeks? a) Yes b) No Is there pain in the jaw when chewing, talking?
  a) Yes b) No Is there pain when chewing, talking?
  a) Yes b) No Is there pain when opening your mouth wide or yawning?
  a) Yes b) No Does biting feel uncomfortable or different from normal?
  a) Yes b) No Have you ever had locking or dislocation of the jaw?
  a) Yes b) No Is there a history of jaw, head or neck injury?
  a) Yes b) No If yes, when? How was it treated? Has he/she ever been treated for a jaw joint disorder?
  a) Yes b) No If so, when? How was it treated? Yes indicates a worse outcome
Detect any negative effects on the TMJ | 3 month
  Clinical examination of the TMJ will be done according to AAPD Guidelines The following questionnaire will be administered to children and parents to detect any negative effects.Does he/she have difficulty opening his/her mouth? a) Yes b) No Do you hear sounds inside your jaw joint? a) Yes b) No Is there pain in the ears or cheeks? a) Yes b) No Is there pain in the jaw when chewing, talking?
  a) Yes b) No Is there pain when chewing, talking?
  a) Yes b) No Is there pain when opening your mouth wide or yawning?
  a) Yes b) No Does biting feel uncomfortable or different from normal?
  a) Yes b) No Have you ever had locking or dislocation of the jaw?
  a) Yes b) No Is there a history of jaw, head or neck injury?
  a) Yes b) No If yes, when? How was it treated? Has he/she ever been treated for a jaw joint disorder?
  a) Yes b) No If so, when? How was it treated? Yes indicates a worse outcome
Detect any negative clinical effects of placing an HTPMC on the masseter muscles. | Baseline
  Masseter muscles will be examined to evaluate the clinical symptoms following placement of an HTPMC on these tissues. American Academy of Pediatric Dentistry Guidelines will be used for the examination The following questionnaire will be administered to children and parents to detect any negative effects.1. The presence of sensitivity, pain or reflected pain on palpation of the masticatory muscles and cervical muscles 0=no pain, 1=palpable pain, and 2=palpebral reflex 2. Pain on palpation of the lateral capsule of the TMJs; 0=no pain, 1=palpable pain, and 2=palpebral reflex 3. Palpation and auscultation for TMJ sounds a)Available b)None 4. Limitation of mandibular movements a)Available b)None 5. Maximum opening: 0=≥35 mm, 1=25-34 mm, 2=<25 mm 6. Deflection during movement: 0=<2mm,1=2-5mm, 2=>5 mm 7.Impaired TMJ function: a)clicking b)deadlock c)luxation 0=no impairment,1=palpable click, 2=audible click, deadlock, or luxation A higher the score, indicates a worse outcome
Detect any negative clinical effects of placing an HTPMC on the masseter muscles. | Immediately after treatment
  Masseter muscles will be examined to evaluate the clinical symptoms following placement of an HTPMC on these tissues. American Academy of Pediatric Dentistry Guidelines will be used for the examination The following questionnaire will be administered to children and parents to detect any negative effects. 1. The presence of sensitivity, pain or reflected pain on palpation of the masticatory muscles and cervical muscles 0=no pain, 1=palpable pain, and 2=palpebral reflex 2. Pain on palpation of the lateral capsule of the TMJs; 0=no pain, 1=palpable pain, and 2=palpebral reflex 3. Palpation and auscultation for TMJ sounds a)Available b)None 4. Limitation of mandibular movements a)Available b)None 5. Maximum opening: 0=≥35 mm, 1=25-34 mm, 2=<25 mm 6. Deflection during movement: 0=<2mm,1=2-5mm, 2=>5 mm 7.Impaired TMJ function: a)clicking b)deadlock c)luxation 0=no impairment,1=palpable click, 2=audible click, deadlock, or luxation A higher the score, indicates a worse outcome
Detect any negative clinical effects of placing an HTPMC on the masseter muscles. | 1 month
  Masseter muscles will be examined to evaluate the clinical symptoms following placement of an HTPMC on these tissues. American Academy of Pediatric Dentistry Guidelines will be used for the examination The following questionnaire will be administered to children and parents to detect any negative effects.1. The presence of sensitivity, pain or reflected pain on palpation of the masticatory muscles and cervical muscles 0=no pain, 1=palpable pain, and 2=palpebral reflex 2. Pain on palpation of the lateral capsule of the TMJs; 0=no pain, 1=palpable pain, and 2=palpebral reflex 3. Palpation and auscultation for TMJ sounds a)Available b)None 4. Limitation of mandibular movements a)Available b)None 5. Maximum opening: 0=≥35 mm, 1=25-34 mm, 2=<25 mm 6. Deflection during movement: 0=<2mm,1=2-5mm, 2=>5 mm 7.Impaired TMJ function: a)clicking b)deadlock c)luxation 0=no impairment,1=palpable click, 2=audible click, deadlock, or luxation A higher the score, indicates a worse outcome
Detect any negative clinical effects of placing an HTPMC on the masseter muscles. | 3 month
  Masseter muscles will be examined to evaluate the clinical symptoms following placement of an HTPMC on these tissues. American Academy of Pediatric Dentistry Guidelines will be used for the examination The following questionnaire will be administered to children and parents to detect any negative effects.1. The presence of sensitivity, pain or reflected pain on palpation of the masticatory muscles and cervical muscles 0=no pain, 1=palpable pain, and 2=palpebral reflex 2. Pain on palpation of the lateral capsule of the TMJs; 0=no pain, 1=palpable pain, and 2=palpebral reflex 3. Palpation and auscultation for TMJ sounds a)Available b)None 4. Limitation of mandibular movements a)Available b)None 5. Maximum opening: 0=≥35 mm, 1=25-34 mm, 2=<25 mm 6. Deflection during movement: 0=<2mm,1=2-5mm, 2=>5 mm 7.Impaired TMJ function: a)clicking b)deadlock c)luxation 0=no impairment,1=palpable click, 2=audible click, deadlock, or luxation A higher the score, indicates a worse outcome
Detect any negative clinical effects of placing an HTPMC on the masseter muscles. | 3 month
  Masseter muscles will be examined to evaluate the clinical symptoms following placement of an HTPMC on these tissues. American Academy of Pediatric Dentistry Guidelines will be used for the examination The following questionnaire will be administered to children and parents to detect any negative effects.1. The presence of sensitivity, pain or reflected pain on palpation of the masticatory muscles and cervical muscles 0=no pain, 1=palpable pain, and 2=palpebral reflex 2. Pain on palpation of the lateral capsule of the TMJs; 0=no pain, 1=palpable pain, and 2=palpebral reflex 3. Palpation and auscultation for TMJ sounds a)Available b)None 4. Limitation of mandibular movements a)Available b)None 5. Maximum opening: 0=≥35 mm, 1=25-34 mm, 2=<25 mm 6. Deflection during movement: 0=<2mm,1=2-5mm, 2=>5 mm 7.Impaired TMJ function: a)clicking b)deadlock c)luxation 0=no impairment,1=palpable click, 2=audible click, deadlock, or luxation A higher the score, indicates a worse outcome.
Evaluate the child's satisfaction with their HTPMC. | 3 Month
  A questionnaire will be carried out through an interview with children to determine what their perception of HTPMC and the procedure is.
  1. I am happy with my fixed tooth
  2. I show my fixed tooth to my friends
  3. I feel happy if people ask to see my fixed tooth
  4. I can eat well with my fixed tooth
  5. My fixed tooth never hurts me
  The scale is 0 (strongly agree) 1 (agree) 2 (no opinion) 3 (disagree) 4 (strongly disagree) A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola INNES, PhD, Study Chair — Cardiff University
Locations (1):
- Melis AKYILDIZ, Efeler, Aydın, Turkey (Türkiye)

REFERENCES:
- [Background] Uribe SE, Innes N, Maldupa I. The global prevalence of early childhood caries: A systematic review with meta-analysis using the WHO diagnostic criteria. Int J Paediatr Dent. 2021 Nov;31(6):817-830. doi: 10.1111/ipd.12783. Epub 2021 Apr 30. PMID 33735529
- [Background] Klingberg G, Broberg AG. Dental fear/anxiety and dental behaviour management problems in children and adolescents: a review of prevalence and concomitant psychological factors. Int J Paediatr Dent. 2007 Nov;17(6):391-406. doi: 10.1111/j.1365-263X.2007.00872.x. PMID 17935593
- [Background] Innes NP, Evans DJ, Stirrups DR. The Hall Technique; a randomized controlled clinical trial of a novel method of managing carious primary molars in general dental practice: acceptability of the technique and outcomes at 23 months. BMC Oral Health. 2007 Dec 20;7:18. doi: 10.1186/1472-6831-7-18. PMID 18096042
- [Background] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395
- [Background] Abu Serdaneh S, AlHalabi M, Kowash M, Macefield V, Khamis AH, Salami A, Hussein I. Hall technique crowns and children's masseter muscle activity: A surface electromyography pilot study. Int J Paediatr Dent. 2020 May;30(3):303-313. doi: 10.1111/ipd.12611. Epub 2020 Jan 24. PMID 31894621
- [Background] Shih YC, Yang R, Zou J. Assessment of occlusion and temporomandibular joint after placing preformed metal crowns on all primary molars in children. Int J Paediatr Dent. 2022 Nov;32(6):915-924. doi: 10.1111/ipd.12970. Epub 2022 May 18. PMID 35484864
- [Background] Elamin F, Abdelazeem N, Salah I, Mirghani Y, Wong F. A randomized clinical trial comparing Hall vs conventional technique in placing preformed metal crowns from Sudan. PLoS One. 2019 Jun 3;14(6):e0217740. doi: 10.1371/journal.pone.0217740. eCollection 2019. PMID 31158253
- [Background] Hesse D, de Araujo MP, Olegario IC, Innes N, Raggio DP, Bonifacio CC. Atraumatic Restorative Treatment compared to the Hall Technique for occluso-proximal cavities in primary molars: study protocol for a randomized controlled trial. Trials. 2016 Mar 31;17:169. doi: 10.1186/s13063-016-1270-z. PMID 27029801